CLINICAL TRIAL: NCT03786341
Title: Kaohsiung Veterans General Hospital , Kaohsiung, Taiwan
Brief Title: Efficacy of a Novel Walking Assist Device With Auxiliary Laser Illuminator on Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Wan-Yun Huang, Department of Physical Medicine and Rehabilitation, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHKS17-CT8-11
Record Dates: First submitted 2018-12-15; First posted 2018-12-26 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: Gait; Stroke; Walking assist device; Auxiliary illuminator; visual feedback
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This was a randomized-prospective study and participants were recruited to each the experimental and the control group equally. Patients in the experimental group (EG) received 30-minutes rehabilitation, consisting of 15 minutes of walking training with laser quad-cane and 15 minutes of traditional physical therapy (such as strengthening and balance training). Patients in the control group (CG) received the same rehabilitation except that the walking training was by conventional strategy without lase quad-cane. The rehabilitation lasted for 4 weeks, twice per week. Gait parameters were measured by Rehab watch as primary outcomes and Berg's balance scale (BBS), timed-up-and-go test (TUG), and Barthel index were used as secondary outcomes. Both the primary and secondary outcomes were measured before the rehabilitation (baseline), 4 weeks (week 4), and 8 weeks (week 8) after the rehabilitation.
Who Masked: Outcomes Assessor
Masking Description: Patients who fulfilled the inclusion and exclusion criteria were randomized (1:1) into two groups, using sequentially numbered, opaque, sealed envelopes (SNOSE) method containing a group assignment number by a person who was not clinically involved in and, therefore, was blinded to this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with auxiliary illuminator (Experimental): the walking training was by conventional strategy with lase quad-cane.
  Interventions: Device: with auxiliary illuminator
- control group (Placebo Comparator): Ambulation training WITHOUT laser quad-cane.
  Interventions: Device: with auxiliary illuminator

INTERVENTIONS:
Device: with auxiliary illuminator — Ambulation training with laser quad-cane for 15 minutes and typical physical therapy with strengthening and balance training for 15 minutes.
  Other Names: control group

SUMMARY:
Many patients after acute stage of stroke present with abnormal gait pattern due to weakness or hypertonicity of the affected limbs.

Ambulation training with the use of visual feedback strategy is one of the promising rehabilitation in patients with chronic stroke.

Walking assist device with auxiliary laser illuminator during ambulation training could correct gait parameters, improve balance and basic activity of daily living among stroke patients.

DETAILED DESCRIPTION:
Facilitation of normal gait is a primary goal of rehabilitation on patients with stroke. The investigators aimed to investigate whether walking assist device with auxiliary lser illuminator (laser quad-cane) providing visual feedback during ambulation could improve parameters of gait cycle and function among patients with chronic stroke.

Methods: This was a randomized-prospective study and participants were recruited to each the experimental and the control group equally. Patients in the experimental group (EG) received 30-minutes rehabilitation, consisting of 15 minutes of walking training with laser quad-cane and 15 minutes of traditional physical therapy (such as strengthening and balance training). Patients in the control group (CG) received the same rehabilitation except that the walking training was by conventional strategy without lase quad-cane. The rehabilitation lasted for 4 weeks, twice per week. Gait parameters were measured by Rehab watch as primary outcomes and Berg's balance scale (BBS), timed-up-and-go test (TUG), and Barthel index were used as secondary outcomes. Both the primary and secondary outcomes were measured before the rehabilitation (baseline), 4 weeks (week 4), and 8 weeks (week 8) after the rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients at subacute (stroke symptoms between three months to one year) or chronic stage (stroke symptoms more than 1 year)
* with hemiplegia
* with sufficient cognition that could follow the instructions and procedure
* walk independently for a distance of more than 20 meters with or without the use of a walking aid.

Exclusion Criteria:

* Stroke patients with other neurological diseases like Parkinsonism,
* Myopathy
* Multiple sclerosis
* Spinal cord injury that might interfere with walking ability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
The change of stride length (meter) of parameters of gait cycle. | The study consisted of a screen visit, a baseline visit and follow-up visits at 4 and 8 weeks after the initiation of the study.
  The primary outcome was the stride length (meter) of parameters of gait cycle. The parameters of gait cycle were measured by a gait analyzer (Reha-Watch1 system; HASOMED1 GmbH, Magdeburg, Germany). Reha-Watch 1 system is based on inertial sensors that allow the quantitative measurement of the important kinematic variables acceleration and angular velocity. The associated software analyzes the sensor signals and calculates temporal (e.g., stride duration, gait phases) and spatial (e.g., stride length, foot angle) parameters on this basis.
The change of cadence(step/min) of parameters of gait cycle | The study consisted of a screen visit, a baseline visit and follow-up visits at 4 and 8 weeks after the initiation of the study.
  The primary outcome was the cadence(step/min) of parameters of gait cycle. The parameters of gait cycle were measured by a gait analyzer (Reha-Watch1 system; HASOMED1 GmbH, Magdeburg, Germany). Reha-Watch 1 system is based on inertial sensors that allow the quantitative measurement of the important kinematic variables acceleration and angular velocity. The associated software analyzes the sensor signals and calculates temporal (e.g., stride duration, gait phases) and spatial (e.g., stride length, foot angle) parameters on this basis.
The change of duration of stance phase(%) of parameters of gait cycle | The study consisted of a screen visit, a baseline visit and follow-up visits at 4 and 8 weeks after the initiation of the study.
  The primary outcome was the duration of stance phase(%) of parameters of gait cycle. The parameters of gait cycle were measured by a gait analyzer (Reha-Watch1 system; HASOMED1 GmbH, Magdeburg, Germany). Reha-Watch 1 system is based on inertial sensors that allow the quantitative measurement of the important kinematic variables acceleration and angular velocity. The associated software analyzes the sensor signals and calculates temporal (e.g., stride duration, gait phases) and spatial (e.g., stride length, foot angle) parameters on this basis.
The change of duration of swing phase(%) of parameters of gait cycle | The study consisted of a screen visit, a baseline visit and follow-up visits at 4 and 8 weeks after the initiation of the study.
  The primary outcome was the duration of swing phase(%) of parameters of gait cycle. The parameters of gait cycle were measured by a gait analyzer (Reha-Watch1 system; HASOMED1 GmbH, Magdeburg, Germany). Reha-Watch 1 system is based on inertial sensors that allow the quantitative measurement of the important kinematic variables acceleration and angular velocity. The associated software analyzes the sensor signals and calculates temporal (e.g., stride duration, gait phases) and spatial (e.g., stride length, foot angle) parameters on this basis.
The change of duration of single support (%) of parameters of gait cycle | The study consisted of a screen visit, a baseline visit and follow-up visits at 4 and 8 weeks after the initiation of the study.
  The primary outcome was the duration of single support (%) of parameters of gait cycle. The parameters of gait cycle were measured by a gait analyzer (Reha-Watch1 system; HASOMED1 GmbH, Magdeburg, Germany). Reha-Watch 1 system is based on inertial sensors that allow the quantitative measurement of the important kinematic variables acceleration and angular velocity. The associated software analyzes the sensor signals and calculates temporal (e.g., stride duration, gait phases) and spatial (e.g., stride length, foot angle) parameters on this basis.
The change of double support (%)during the gait cycle | The study consisted of a screen visit, a baseline visit and follow-up visits at 4 and 8 weeks after the initiation of the study.
  The primary outcome was the double support (%)during the gait cycle. The parameters of gait cycle were measured by a gait analyzer (Reha-Watch1 system; HASOMED1 GmbH, Magdeburg, Germany). Reha-Watch 1 system is based on inertial sensors that allow the quantitative measurement of the important kinematic variables acceleration and angular velocity. The associated software analyzes the sensor signals and calculates temporal (e.g., stride duration, gait phases) and spatial (e.g., stride length, foot angle) parameters on this basis.
The change ofangle between toes and the ground at the time of toe-off during a gait cycle (toe-off angle) | The study consisted of a screen visit, a baseline visit and follow-up visits at 4 and 8 weeks after the initiation of the study.
  The primary outcome was the angle between toes and the ground at the time of toe-off during a gait cycle (toe-off angle). The parameters of gait cycle were measured by a gait analyzer (Reha-Watch1 system; HASOMED1 GmbH, Magdeburg, Germany). Reha-Watch 1 system is based on inertial sensors that allow the quantitative measurement of the important kinematic variables acceleration and angular velocity. The associated software analyzes the sensor signals and calculates temporal (e.g., stride duration, gait phases) and spatial (e.g., stride length, foot angle) parameters on this basis.
The change ofangle between calcaneus and the ground at the time of heel-strike during a gait cycle (heel-strike angle) | The study consisted of a screen visit, a baseline visit and follow-up visits at 4 and 8 weeks after the initiation of the study.
  The primary outcome was the angle between calcaneus and the ground at the time of heel-strike during a gait cycle (heel-strike angle). The parameters of gait cycle were measured by a gait analyzer (Reha-Watch1 system; HASOMED1 GmbH, Magdeburg, Germany). Reha-Watch 1 system is based on inertial sensors that allow the quantitative measurement of the important kinematic variables acceleration and angular velocity. The associated software analyzes the sensor signals and calculates temporal (e.g., stride duration, gait phases) and spatial (e.g., stride length, foot angle) parameters on this basis.

SECONDARY OUTCOMES:
The Berg balance scale (BBS) | The study consisted of a screen visit, a baseline visit and follow-up visits at 4 and 8 weeks after the initiation of the study.
  The Berg balance scale (BBS) is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. It is used to objectively determine a patient's ability to safely balance during a series of predetermined tasks. The higher the score means the better ability to maintain the balance. A score of less than 45 indicates individuals may be at greater risk of falling. Studies of various populations and stroke patients have shown high intra-rater and inter-rater reliability (intraclass correlation coefficient [ICC]=0.98 and 0.97, respectively). BBS has been reported that in the elderly population a change of 4 points is needed to be 95% confident that true change has occurred if a patient scores within 45-56 initially, 5 points if they score within 35-44, 7 points if they score within 25-34 and, finally, 5 points if their initial score is within 0-24 on the Berg Balance Scale.
Barthel index (BI) | The study consisted of a screen visit, a baseline visit and follow-up visits at 4 and 8 weeks after the initiation of the study.
  Barthel index (BI) measures the degree of assistance required by an individual on 10 items of mobility and self-care Activity of daily living, including feeding, dressing, grooming, bathing, bowels, bladder, toilet use, transfers, mobility, and stairs. The total scores ranges from 0 to 100. The higher the score means the better of the function. BI has been shown to have portability and has been used in 16 major diagnostic conditions. Studies has demonstrated high inter-rater reliability (0.95) and test-retest reliability (0.89) as well as high correlations (0.74-0.8) with different physical disabilities.
Timed up and go test (TUG) | The study consisted of a screen visit, a baseline visit and follow-up visits at 4 and 8 weeks after the initiation of the study.
  Timed up and go test (TUG) is designed for determining fall risk and measuring the progress of balance, sit to stand, and walking. To perform the test, participant starts in a seated position (50 cm from the floor), stands up upon therapist's command to walk 3 meters, then turn around, walk back to the chair and sit down. The time stops when the patient is seated. If a community dwelling older adults takes 14 seconds or longer, the risk for falling is high. The TUG showed excellent reliability (ICC>0.95) in chronic stroke patients.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Te Hsu, MD., Study Director — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital ,, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
to publish the journal